CLINICAL TRIAL: NCT04466098
Title: Multi-center, Randomized, Placebo Controlled, Interventional Phase 2A Clinical Trial Evaluating the Safety and Potential Efficacy of Multiple Dosing of Mesenchymal Stromal Cells in Patients With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-Cov-2)
Brief Title: Multiple Dosing of Mesenchymal Stromal Cells in Patients With ARDS (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020LS075; MT2020-12 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2020-07-08; First posted 2020-07-10 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Acute Respiratory Distress Syndrome; ARDS (Moderate or Severe); COVID-19 Pneumonia
Keywords: cytokine storm; Mesenchymal Stem Cells; SARS-CoV-2; COVID-19; Mesenchymal Stromal Cells; MSC
MeSH Terms: conditions — Respiratory Distress Syndrome; Lymphoma, Follicular; Cytokine Release Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: This is a randomized (2:1 ratio) placebo controlled trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be randomly assigned (2:1) to receive either 300 × 10^6 MSC or vehicle placebo control. Randomization will be stratified by risk (high versus standard risk based on the presence of preexisting co-morbidities), using permuted block sizes of 3. The allocation sequence will be accessed by each cell processing laboratory through ONCORE. Personnel in the cell processing laboratories are not masked to the treatment group, but patients, clinical staff, and investigators will be unaware of treatment assignment. To maintain masking of the investigators and clinicians, bags containing the study products and intravenous tubing had opaque coverings applied in the cell laboratories.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mesenchymal Stromal Cells (Experimental): Three fixed doses of MSC approximately 48 hours apart.
  Interventions: Biological: Mesenchymal stromal cells
- Placebo (Placebo Comparator): Three fixed doses of placebo control approximately 48 hours apart.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Mesenchymal stromal cells — Thawed product containing MSC(300x10^6) in DMSO resuspended 1:1 with Dextran 40 + 5% human serum albumin [total volume 60 mL]
  Other Names: MSC
  Arms: Mesenchymal Stromal Cells
Other: Placebo — Dextran 40 + 5% human serum albumin [total volume 60 mL]
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, placebo controlled, interventional phase 2A trial to evaluate the safety profile and potential efficacy of multi-dosing of mesenchymal stromal cells (MSC) for patients with SARS-CoV-2 associated Acute Respiratory Distress Syndrome (ARDS). After informed consent, treatment assignment will be made by computer-generated randomization to administer either MSC or vehicle placebo control with a 2:1 allocation to the MSC: placebo arm.

DETAILED DESCRIPTION:
MSCs are adult, non-hematopoietic precursor cells derived from a variety of tissues (e.g., bone marrow, adipose tissue, and placenta) and have been used as therapy in multiple conditions, especially in immune-mediated inflammatory diseases, such as graft versus-host disease (GVHD) and systemic lupus erythematosus (SLE) with evidence of benefit.

In preclinical models, MSC are effective in ameliorating acute lung injury due to their ability to secrete paracrine factors that regulate lung endothelial and epithelial permeability, including growth factors, anti-inflammatory cytokines, and antimicrobial peptides. Based on the promising pre-clinical preliminary data and intriguing results in patients with COVID-19 associated pneumonia and ARDS as well as an established safety profile of MSC generally and in ARDS in particular, the researchers propose multiple dosing of MSCs as a study treatment to ameliorate the severity and duration of SARS-CoV-2 associated pneumonia and ARDS potentially improve survival.

Patients will receive study agent (MSC or placebo) within 48 hours of enrollment. Three doses will be administered unless a severe infusion adverse event occurs that is related to the MSC infusion. Doses will be repeated approximately every 48-72 hours with the aim of completing 3 doses within 7 days of the first dose. All patients will receive standard of care treatments for ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Meets 'Berlin Criteria' for diagnosis of moderate to severe ARDS for a minimum of 4 hours
* Less than 48 hours on a ventilator after meeting criteria for diagnosis of ARDS
* SARS-CoV-2 (proven by RT-PCR assay) with radiographic infiltrates
* PaO2/FiO2 < 250
* Positive end-expiratory airway pressure (PEEP) >5 cm H20
* Elevated C-reactive protein (above laboratory upper limit of normal)
* Meets organ function requirements, including left ventricular ejection fraction (LVEF) >35% ( as defined below)
* Off other investigational agents directed against inflammatory cytokines 48 hours prior to enrollment; agents directed against the replication of SARS-CoV-2 [e.g., Remdesivir] are permitted
* Voluntary informed consent in person or virtually by the patient or patient surrogate considering the face to face limitations during the COVID-19 pandemic and, given the nature of the study population, which frequently requires mechanical ventilation with sedation, surrogate consent will likely occur in a substantial proportion of the study population (this will remain a valid consent until the patient is fully alert, and aware, and can provide a second consent to continue participation in the study).
* Adequate organ function is defined as:

  * Renal: Calculated estimated glomerular filtration rate >30 mL/min/1.73 m2 (on chemistry panel)
  * Hepatic: Bilirubin <3x upper limit of normal (ULN) and AST, ALT and alkaline phosphatase <5x ULN
  * Cardiac: Absence of uncontrolled arrhythmia and LVEF >35%

Exclusion Criteria:

* Ventilator support of FiO2 >0·8 or PEEP >20 cm H2O and ongoing use of more than two vasopressors for 2 or more hours with any agent at doses shown below in the supine position.

  * Norepinephrine >12 μg/min or 0.2 μg/kg per min
  * Phenylephrine >150 μg/min or 3 μg/kg per min
  * Epinephrine >10 ug/min or 0.2 μg/kg per min
  * Vasopressin >0.04 units/min
* Concurrent use of other investigational agents specifically for treatment of ARDS or inflammatory cytokines. (Note: Agents established to be efficacious and/or those used outside of formal trials are permitted as supportive data emerge)
* Known ineligibility for use of a ventilator for a minimum of 7 days, as judged by the institution's Triage Team
* Known allergy to MSC components: fetal calf serum, human albumin or DMSO
* Active invasive malignant disease requiring chemotherapy/radiation
* Other concurrent life-threatening disease (life expectancy <6 months) or eligible for hospice care
* Known history of HIV infection on active treatment
* Females who are pregnant or breastfeeding
* Current mean arterial pressure (MAP) <60 mmHg while on 2 or more vasopressors at above doses for more than 2 hours
* History of any significant cardiac (myocardial infarction within 12 months of screening visit or unstable angina), chronic ongoing hepatic, or renal disease (grade 3 or higher); diagnosis of congestive heart failure with hypoxemia primarily due to decompensated heart failure; diagnosis of severe chronic obstructive pulmonary disease (COPD) or interstitial lung disease requiring supplemental oxygen at home
* Concurrent diagnosis of diffuse alveolar hemorrhage
* Requiring continuous dialysis (unable to stop dialysis during study agent infusion)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ingbar, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - University of Pittsburgh, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mesenchymal Stromal Cells | Placebo
Started | 6 | 2
Completed | 3 | 0
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesenchymal Stromal Cells | Placebo | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade 3-5 Infusional Toxicities and Predefined Hemodynamic or Respiratory Adverse Events Related to the Infusion of MSC
Time Frame: Within 6 hours of the start of the infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
Participants | 0 | 0

2. Secondary Outcome: Change in Biomarkers of Inflammation From Day 0 to Day 7
Description: Mean (SD) represents the change on day 7 after treatment compared to pretreatment value for each biomarker of inflammation. (IL-1, IL-6, IL-8 and TNFa) Measured in pg/mL.
Time Frame: Day 7 after first infusion
Population: One participant in 'Mesenchymal Stromal Cells' arm unable to be evaluated.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
pg/mL
  Change in IL-1 | 0 (0.55) | 0.4 (0.99)
  Change in IL-6: number analyzed (Participants) | 5 | 2
  Change in IL-6 | -61 (190) | 102 (75)
  Change in TNFa: number analyzed (Participants) | 5 | 2
  Change in TNFa | 0 (12) | 2 (2)
  Change in IL-8: number analyzed (Participants) | 5 | 2
  Change in IL-8 | 6 (53) | 145 (33)

3. Secondary Outcome: Trend Changes in PaO2:FiO2 Ratio
Description: Trend change was determined by evaluating PaO2:FiO2 ratios at prespecified time points and determining the slope of the line of best fit across data points for each patient, followed by taking the mean and SD across patients in each treatment group. Negative and positive slopes indicating decreasing or increasing values over time, respectively.
Time Frame: On the day of screening and on days 3, 7 and 14 after first infusion
Measure: Mean (Standard Deviation); unit: ratio/day
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
ratio/day | -7 (8) | 8 (7)

4. Secondary Outcome: Trend Changes in Mean Airway Pressure
Description: Trend change was determined by evaluating mean airway pressure values at prespecified time points and determining the slope of the line of best fit across data points for each patient, followed by taking the mean and SD across patients in each treatment group. Negative and positive slopes indicating decreasing or increasing values over time, respectively.
Time Frame: On the day of screening and on days 3, 7 and 14 after first infusion
Measure: Mean (Standard Deviation); unit: ratio/day
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
ratio/day | -2.7 (6) | 0.3 (0.4)

5. Secondary Outcome: Trend Changes in Peak Pressure
Description: Trend change was determined by evaluating peak pressure values at prespecified time points and determining the slope of the line of best fit across data points for each patient, followed by taking the mean and SD across patients in each treatment group. Negative and positive slopes indicating decreasing or increasing values over time, respectively.
Time Frame: On the day of screening and on days 3, 7 and 14 after first infusion
Measure: Mean (Standard Deviation); unit: ratio/day
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
ratio/day | -0.28 (1.51) | 0.19 (0.45)

6. Secondary Outcome: Trend Changes in Plateau Pressure
Description: Trend change was determined by evaluating plateau pressure values at prespecified time points and determining the slope of the line of best fit across data points for each patient, followed by taking the mean and SD across patients in each treatment group. Negative and positive slopes indicating decreasing or increasing values over time, respectively.
Time Frame: On the day of screening (baseline) and on days 3, 7 and 14 after first infusion
Measure: Mean (Standard Deviation); unit: ratio/day
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
ratio/day | 0.08 (2.91) | 0.38 (0.71)

7. Secondary Outcome: Trend Changes in Positive End-expiratory Airway Pressure (PEEP)
Description: Trend change was determined by evaluating Positive end-expiratory airway pressure (PEEP) values at prespecified time points and determining the slope of the line of best fit across data points for each patient, followed by taking the mean and SD across patients in each treatment group. Negative and positive slopes indicating decreasing or increasing values over time, respectively.
Time Frame: On the day of screening and on days 3, 7 and 14 after first infusion
Measure: Mean (Standard Deviation); unit: ratio/day
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
ratio/day | -0.68 (0.90) | 0.14 (0.28)

8. Secondary Outcome: Incidence of Mortality
Time Frame: 50 days after first infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
Participants | 2 | 1

9. Secondary Outcome: Number of ICU-free Days
Time Frame: 28 days after first infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
Participants
  0 days | 3 | 2
  7 days | 1 | 0
  18 days | 1 | 0
  22 days | 1 | 0

10. Secondary Outcome: Number of Days Alive and Ventilator Free
Time Frame: 28 days after first infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
Participants
  0 days | 3 | 1
  1 day | 0 | 1
  4 days | 1 | 0
  23 days | 1 | 0
  24 days | 1 | 0

11. Secondary Outcome: Change in Acute Lung Injury (ALI) Score 2
Description: Acute Lung Injury Score is a composite 4 point scoring system validated by the NHLBI ARDS Network that considers PaO2/FiO2, the level of positive end-expiratory airway pressure, respiratory compliance, and the extent of pulmonary infiltrates on the chest radiograph. Each criterion is scored from 0-4 based on the severity of the condition. The final score is calculated by dividing the total score by the number of criteria used. A score of 0 indicates no lung injury, and a score over 2.5 indicates Acute respiratory distress syndrome (ARDS). The scoring ranges from 0 to a maximum score of 3.
Time Frame: Baseline and Day 28 after first infusion
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 3 | 1
Scores on a scale | -0.25 (0.43) | -1.5 (0)

12. Secondary Outcome: Incidence of Serious Adverse Events
Time Frame: 28 days after first infusion
Measure: Number; unit: Participants
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
Participants | 2 | 1

13. Secondary Outcome: Number of Days Alive Off Supplemental Oxygen
Time Frame: 100 days after first infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stromal Cells | Placebo
Number analyzed (Participants) | 6 | 2
Participants
  0 days | 2 | 1
  10 days | 1 | 0
  53 days | 0 | 1
  61 days | 1 | 0
  87 days | 1 | 0
  88 days | 1 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Mesenchymal Stromal Cells | Placebo
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/2
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/2
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesenchymal Stromal Cells (N=6) | Placebo (N=2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesenchymal Stromal Cells (N=6) | Placebo (N=2)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 2 (2) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 3 (3) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT04466098/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT04466098/ICF_001.pdf